CLINICAL TRIAL: NCT05602116
Title: Effect of Adipose Tissue Derived Mesenchymal Stromal Cells on Autism and Leaky Gut Syndrome. A Phase I Pilot Study.
Brief Title: ASC - Autism Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cell to Cure ApS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASC II
Record Dates: First submitted 2022-09-23; First posted 2022-11-01 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder; Gastrointestinal Dysfunction; Leaky Gut Syndrome; Mesenchymal Stromal Cells; Inflammatory Bowel Diseases
Keywords: Gastrointestinal microbiota; Gut-brain axis; Immunomodulation
MeSH Terms: conditions — Autism Spectrum Disorder; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Open dose titrating with two groups in extension of each other (thus not categorically parallel).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 x 1000000 C2C_ASCs/kg body weight (Experimental): Trial participant 1 - 5 will be treated with 1 x 1000000 C2C_ASCs/kg body weight
  Interventions: Drug: Adipose tissue derived mesenchymal stromal/stem cells (Cell2Cure®)
- 2 x 1000000 C2C_ASCs/kg body weight (Experimental): Trial participant 6 - 10 will be treated with 2 x 1000000 C2C_ASCs/kg body weight
  Interventions: Drug: Adipose tissue derived mesenchymal stromal/stem cells (Cell2Cure®)

INTERVENTIONS:
Drug: Adipose tissue derived mesenchymal stromal/stem cells (Cell2Cure®) — The Investigational Product is a C2C_ASC cell product (Cell2Cure®, Cell2Cure Aps, Denmark).
  C2C_ASC is an advanced therapy investigational medicinal product (ATIMP) manufactured from abdominal adipose tissue derived mesenchymal stromal cells (ASC) from healthy donors. C2C_ASC is aseptically procured and manufactured according to tissue law and GMP by Cell2Cure ApS or Cardiology Stem Cell Center, Rigshospitalet, Copenhagen, Denmark, using manual isolation of cells from abdominal fat tissue, xeno-free cell expansion in automated closed bioreactor systems and cryopreservation of the final product.
  The active substance is the in vitro expanded ASCs. The final product, C2C_ASC, is provided as a cryopreserved suspension of 50 million ASCs per ml with a total volume of 1,3 ml per vial. The excipient is CryoStor10 (Biolife Solutions), holding 10% DMSO.

SUMMARY:
The ASC - Autism Pilot Study is a single center randomized open dose titrating phase I clinical intervention pilot trial with the aim of investigating safety and treatment effect of an allogeneic adipose tissue derived mesenchymal stromal cell product (C2C_ASC) in children with autism spectrum disorder (ASD) and gastrointestinal symptoms.

DETAILED DESCRIPTION:
The ASC - Autism Pilot Study will be performed at the Child and Adolescent Psychiatry, Aalborg University Hospital, Denmark. 10 children aged 6-14 years with ASD and gastrointestinal symptoms will be enrolled through the Child and Adolescent Psychiatry, Psychiatry Clinic South, Aalborg University Hospital, Denmark.

The participants will randomly be divied into two treatment groups:

1. participant 1-5 will be treated with 1 x 1000000 C2C_ASCs/kg body weight
2. participant 6-10 will be treated with 2 x 1000000 C2C_ASCs/kg body weight

C2C_ASC treatment:

The C2C_ASCs product will be diluted in 50 ml isotonic saline and infused in an arm vein within 15 min. In both groups there will for each participant be a week observation for SAE's related to the cell treatment before the next participant will be treated, if no SAE's have been detected.

The investigators hypothesize that the connection between gastrointestinal symptoms/leaky gut syndrome, increase local gastrointestinal and systemic elevated immunological and inflammatory activity, bacterial toxins in the blood and symptoms of ASD in children with symptoms of leaky gut syndrome can be reduced or normalized by modulating the immunological activity and inflammation by treatment with mesenchymal stromal cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder.
* Ongoing gastrointestinal symptoms or previous gastrointestinal symptoms which disappeared or were reduced after dietary changes.
* Age 6 to 14 years.

Exclusion Criteria:

* Known genetic syndrome or pathogenic mutation or copy number variation associated with autism spectrum disorder.
* Known CNS-infection (now or previously) and/or HIV positivity.
* Primary immunodeficiency disorder or autoimmune cytopenia.
* Current treatment with cytotoxic drugs or systemic administered glucocorticoids and/or immunosuppressive therapy or other antiinflammatory medication (except nonsteroidal anti-inflammatory drugs).
* Epilepsy or known seizure disorder (now or previously).

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Safety of C2C_ASC (Adverse Events) | 12 weeks
  Safety of C2C_ASC within the 12 weeks follow-up period: Adverse event (AE), serious adverse event (SAE), suspected unexpected serious adverse reaction (SUSAR) and development safety update report (DSUR).

SECONDARY OUTCOMES:
Changes in autism spectrum disorder | 12 weeks
  Difference from baseline to follow-up within the group treated with C2C_ASC:
  Changes in autism spectrum disorder score test (questionnaire).
  [Raw scores converting to standard scores and then generates five major domain composite scores: communication, daily living skills, socialization, adaptive behavior composite and motor. For these domains a standard score of 100 is the mean with a standard deviation of 15. This means that a score of 100 is similar to the typical population of the same age. Scores in the range of 86 and above are considered adequate. Scores in the range of 85 and below indicates a significant skill deficit when comparing with the typical population of the same age.
  High scores: standard scores of 130-140 Moderately high scores: standard scores of 115-129 Adequate scores: standard scores of 86-114 Moderately low scores: standard scores of 71-85 Low scores: standard scores of 20-70]
Changes in gastrointestinal symptoms | 12 weeks
  Difference from baseline to follow-up within the group treated with C2C_ASC:
  Changes in The Infant Gastrointestinal Symptom Questionnaire (questionnaire).
  [A 0-100 scale where higher scores indicate better irritable bowel syndrome specific quality of life.]

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kastrup, Study Director — Cell to Cure ApS
Locations (1):
- Department of Child and Adolescent Psychiatry, Psychiatry Clinic South, Aalborg University Hospital, Denmark, Aalborg, Denmark